CLINICAL TRIAL: NCT01063439
Title: Busulfan, Etoposide, Cytarabine and Melphalan (BuEAM) as a Conditioning for Autologous Stem Cell Transplantation in Patients With Diffuse Large B Cell Lymphoma (DLCBL) Previously Treated With Rituximab Based Regimen
Brief Title: BuEAM Conditioning for Autologous Stem Cell Transplantation (ASCT) to Treat Diffuse Large B Cell Lymphoma (DLCBL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Won Sik Lee, Inje University Busan Paik Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BuEAM-DLBCL
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-08

CONDITIONS: Non Hodgkin's Lymphoma
Keywords: DLBCL; NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Busulfan; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BuEAM: Experimental (Experimental): BuEAM: Experimental Busulfan 3.2 mg/kg/d for 2 days, etoposide 400 mg/m2/d for 2 days, cytarabine 1 g/m2 for 2 days, and melphalan 140 mg/m2 for 1 day Intervention: Drug: Busulfan, etoposide, cytarabine, and melphalan
  Interventions: Drug: Busulfan, Etoposide, Cytarabine, Melphalan

INTERVENTIONS:
Drug: Busulfan, Etoposide, Cytarabine, Melphalan — Busulfan 3.2 mg/kg/d for 2 days Etoposide 400 mg/m2/d for 2days Cytarabine 1 g/m2 for 2 days Melphalan 140 mg/m2 for 1 day
  Other Names: BuEAM conditioning

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of busulfan, etoposide, cytarabine and melphalan (BuEAM) including intravenous busulfan instead of BCNU of standard BEAM as a conditioning for autologous stem cell transplantation in patients with NHL.

DETAILED DESCRIPTION:
Among the high-dose conditioning regimens commonly used in patients with NHL are BEAM (BCNU, etoposide, cytarabine, and melphalan), BEAC (BCNU, etoposide, cytarabine, and cyclophosphamide), CBV (cyclophosphamide, carmustine, etoposide), and combination regimen with total body irradiation. Three-year progression free survival of patients with NHL received above high-dose chemotherapy followed by autologous stem cell rescue was reported as 40-50%, which is still unsatisfactory.

Busulfan (Bu)-based preparative regimens, which are commonly used with allogeneic SCT have also been studied with ASCT for lymphomas.

The development of intravenous busulfan achieved 100% bioavailability bypassing the oral route and increased safety and reliability of generating therapeutic busulfan levels, maximizing efficacy.

Recently, one prospective study showed that a combination conditioning regimen of i.v. busulfan, cyclophosphamide, etoposide was found to be well tolerated and seemed to be effective in patients with aggressive NHL.

Another prospective study for multiple myeloma patients showed that i.v. busulfan and melphalan conditioning regimen made no grade 3-4 non-hematological complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a high-intermediate/high risk international prognostic index at a diagnosis or with salvage chemotherapy-sensitive relapse/refractory non Hodgkin's lymphoma
* Patients with histologically confirmed diffuse large B cell lymphoma at diagnosis
* Patients treated with rituximab based regimen previously
* Patients who have not received therapy with high-dose chemotherapy and stem cell transplantation
* Life expectation of at least 3 months
* ECOG performance status ≤ 2 (See Appendix II)
* Adequate hepatic function (serum bilirubin less than 2.0 mg/dL, AST and ALT less than three times the upper normal limit)
* Adequate renal function (serum creatinine less than 2.0 mg/dL).
* Adequate cardiac function (ejection fraction ≥ 45% on MUGA scan or echocardiogram).
* Adequate bone marrow function (ANC ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3).
* All patients are fully informed about the nature and purpose of this study and informed consent should be given before the start of treatment. All patients should fully understand the right of trial abandon without any disadvantage

Exclusion Criteria:

* Patients with central nervous system involvement of lymphoma
* Patients positive for human immunodeficiency virus
* Pregnant or breast feeding woman
* Young woman without pregnancy test prior to treatment or pregnancy test reveals positive.
* Young woman without a reliable and proper contraceptive method
* Man being not willing to contraception
* Concurrent history of neoplasm other than NHL with life expectancy less than 3 months (except for curatively treated non-melanoma skin cancer or in-situ uterine cervix cancer).
* History of clinically significant cardiac dysfunction (e.g. congestive heart failure, symptomatic coronary artery disease, medically uncontrolled arrhythmia) or myocardial infarction within 12 months
* A psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible.
* Significant infection or uncontrolled bleeding
* Enrollment of other clinical trials within 4 weeks prior to treatment
* Any preexisting medical condition of sufficient severity to prevent full compliance with the study
* Patient being not willing to or unable to obey study protocol

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-08 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | three year

SECONDARY OUTCOMES:
overall survival | three year
Response rate according to the International Working Group criteria | after 2 month
Adverse events | From start of conditioning to discharge
•Pharmacogenetic study | After 3 years
  Pharmacogenetic study for predictive or prognostic markers using blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Won Sik Lee, Dr. PhD., Principal Investigator — Inje University
Locations (5):
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan, Busan
  - Asan Medical Center, University of Ulsan, Seoul
  - Seoul National University Hospital, Seoul
  - Yeonsei University Hospital, Seoul
  - Ulsan University Hospital, Ulsan